CLINICAL TRIAL: NCT07255417
Title: The Effect of Visualized Meditation on Anxiety, Pain, and Comfort in Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tuğba Albayram, Research Assistant Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/489
Record Dates: First submitted 2025-11-15; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Colonoscopy; Pain Management; Comfort; Randomised Controlled Trial
Keywords: Colonoscopy; Visualized meditation; Pain; Comfort; Randomized controlled trial
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualized meditation group (Active Comparator): In the study, the experimental group will listen to visualized meditation sessions daily, morning and evening, for three days before the colonoscopy. On the morning of the colonoscopy, patients will be administered a personal information form, STAI1-2, pain scale, and comfort scale. After the procedure, the patients will be taken to the recovery area and will be administered the STAI1-2, pain scale, and comfort scale again.
  Interventions: Other: Visualized meditation group
- Control group (No Intervention): In the study, the control group will be administered a personal information form, STAI1-2, pain scale, and comfort scale on the morning of the colonoscopy. After the procedure, the patients will be taken to the recovery area and the STAI1-2, pain scale, and comfort scale will be administered again. The control group will receive standard clinical care procedures.

INTERVENTIONS:
Other: Visualized meditation group — In the study, the experimental group will listen to visualized meditation sessions daily, morning and evening, for three days before the colonoscopy. On the morning of the colonoscopy, patients will be administered a personal information form, STAI1-2, pain scale, and comfort scale. After the procedure, the patients will be taken to the recovery area and will be administered the STAI1-2, pain scale, and comfort scale again.
  Arms: Visualized meditation group

SUMMARY:
Colonoscopy is one of the most frequently performed procedures for the early diagnosis and treatment of intestinal diseases and plays a crucial role in the diagnosis and treatment of lower gastrointestinal disorders. However, for many patients, colonoscopy is considered an invasive, highly painful, and extremely uncomfortable procedure. Furthermore, the anxiety and fear felt before the procedure can affect patients in many ways. These negative feelings can disrupt patient comfort and cause the pain to become even more severe.

DETAILED DESCRIPTION:
Meditation and visualization exercises have been found to alter an individual's mood and perception. Recent neuroscience literature suggests that meditation practices alter brain chemistry, structure, and function more permanently. Meditation facilitates increased selective attention, which increases the ability to silence unwanted outcomes while focusing on a specific outcome, and reduces activity in the amygdala, which is associated with the production of fear and anxiety. Guided meditation with background music is effective in increasing attention, reducing stress, and therefore improving mental health. Visualization is the conscious control of mental imagery. Imagery often plays a fundamental role not only in experiencing reality but also in creating it. In this context, it can be argued that visualized meditation may also allow for the reshaping of perceived reality, such as anxiety and pain, and reduce their negative effects on the patient. This study was conducted to determine the effects of visualized meditation on anxiety, pain, and comfort in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18, with no hearing impairment,
* Submitting a colonoscopy for the first time,
* Not diagnosed with a psychiatric disorder and therefore not taking medication,
* Willing to participate in the study

Exclusion Criteria:

* Patients who refused to participate in the study, underwent a colonoscopy for biopsy, or underwent deep sedation.
* Patients who volunteered to participate and then wished to withdraw from the study at any stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
VAS Pain and Comfort Scale | From enrollment to the end of treatment at 4 months
  This scale was developed by Price and colleagues (1983). It is used to measure subjective pain and comfort levels. The scale is represented by a 10-cm line representing the lowest and highest pain scores (0: no pain/discomfort, 10: most intolerable pain/discomfort).
The State Trait Anxiety Inventory (STAI) | From enrollment to the end of treatment at 4 months
  The State Trait Anxiety Inventory (STAI), developed by Spielberger et al. in 1964, will be used to measure anxiety in this study. The scale has two dimensions: the STAI-S, which measures state anxiety, and the STAI-T, which measures trait anxiety. The STAI-S and STAI-T each consist of 20 items. Items 1-40 on the scale measure anxiety in four ways. The lowest score for both dimensions of the scale is 20, and the highest score is 80. As the score increases, the level of anxiety also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.